CLINICAL TRIAL: NCT06421090
Title: Safety and Feasibility of Transauricular Vagus Nerve Stimulation in Improving Postoperative Delirium in Elderly Patients: a Randomized Controlled Study
Brief Title: Transauricular Vagal Nerve Stimulation Improves Postoperative Delirium in Elderly Patients
Acronym: Vnstar-IIa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, professor, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VNS20240510IIa
Record Dates: First submitted 2024-05-10; First posted 2024-05-20 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Vagus Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transauricular Vagal Nerve Stimulation (Active Comparator)
  Interventions: Device: Transauricular Vagal Nerve Stimulation
- Transauricular Vagal Nerve sham Stimulation (Sham Comparator)
  Interventions: Device: Transauricular Vagal Nerve Stimulation

INTERVENTIONS:
Device: Transauricular Vagal Nerve Stimulation — Transauricular vagal nerve stimulation，Intervention group25Hz，Control group1Hz

SUMMARY:
To investigate the efficacy and safety of perioperative Transauricular vagal nerve stimulation in improving Postoperative Delirium in elderly patients undergoing elective surgery Lay the groundwork for a Phase III study.

DETAILED DESCRIPTION:
This study aims to conduct a prospective, randomized controlled clinical trial on the preventive use of Transauricular vagal nerve stimulation(taVNS) to improve the incidence of Postoperative Delirium(POD) in elderly patients undergoing anesthesia surgery. The intervention group will receive taVNS, while the control group will only wear a taVNS stimulator without current stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Age≥65 years
* Expected operation time≥ 2 hours
* Postoperative hospital stay≥ 4 days
* Sign the informed consent form

Exclusion Criteria:

* Neurosurgery or cardiac surgery
* Emergency surgery within 6 hours of admission
* End-stage disease with an expected survival of < 3 months
* Preoperative severe cognitive dysfunction affected perioperative cognitive function assessment
* Severe sinus bradycardia, AVB of degree II and above, pacemaker placement

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-05-21 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TaVNS tolerance | 1-5 days after surgery
  The proportion of subjects who completed all the expected interventions
Incidence of adverse events | At discharge，an average of 2 weeks
  Myocardial infarction, cardiac arrest, pulmonary embolism, infection, etc

SECONDARY OUTCOMES:
Incidence of POD at discharge or within 5 days postoperatively | At discharge or within 5 days postoperatively
  POD assessment was performed using the 3D-CAM scale estimate. Assessed 2 times daily until postoperative day 5 or hospital discharge.
Incidence of cognitive decline | Day 1 before surgery, day 5 after surgery, day 90 after surgery
  The MMSE scale and MoCA scale was used for evaluation
All-cause mortality | on the 90 days
Postoperative pain | 1-5 days after surgery
  VAS score
Time of anesthesia recovery | Within 2 hours after the end of the surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No